CLINICAL TRIAL: NCT06154694
Title: In-vivo Evaluation of Glenohumeral Joint Contact Patterns in Osteoarthritic Glenoids
Brief Title: Glenohumeral Joint Contract Patterns in Osteoarthritic Glenoids
Acronym: TSA
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64986
Record Dates: First submitted 2023-10-31; First posted 2023-12-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis of Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Shoulder osteoarthritis patients: Patients with glenohumeral osteoarthritis
  Interventions: Radiation: Stereo Radiographic EOS Measurements
- Healthy control: Healthy adult volunteers with no history of shoulder pain or trauma
  Interventions: Radiation: Stereo Radiographic EOS Measurements

INTERVENTIONS:
Radiation: Stereo Radiographic EOS Measurements — Healthy control will undergo a stereo radiographic EOS exam with their arm in various positions.
  1. Relaxed standing (0 degree of abduction)
  2. 45 degree of abduction in the coronal plane
  3. 90 degree of abduction in the coronal plane
  4. 120 degree of abduction in the coronal plane
  5. 45 degree anterior flexion in the sagittal plane
  6. 90 degree anterior flexion in the sagittal plane
  7. 120 degree of anterior flexion in the sagittal plane
  8. 45 degree extension in the sagittal plane

SUMMARY:
Shoulder osteoarthritis (OA) is a frequent problem in our aging population and is believed to occur in up to 20% of the population. Different types of glenoid morphology are associated with shoulder OA, depending on the amount and localization of the glenoid erosion as well as the amount and direction of Humeral Head Migration.

Total shoulder arthroplasty (TSA) has been shown to relieve the pain and improve joint function of patients with OA. However, several complications such as component loosening and polyethylene damage has been reported and it has been revealed that 7.3% of glenoids may show signs of asymptomatic radiographic loosening annually after primary anatomic TSA. The mechanism of such fixation failure is still unclear.

The main goal of this study is evaluating in-vivo glenohumeral contact patterns in patients with osteoarthritic glenoids before and after TSA, to unravel the high rate of glenoid component loosening.

DETAILED DESCRIPTION:
Shoulder osteoarthritis (OA) is a frequent problem in our aging population and is believed to occur in up to 20% of the population. OA leads to pain, restriction of movement and functional disability. Furthermore, chronic instability, characterized by humeral head migration (HHM), and pathologic changes of the glenoid bone, i.e. glenoid erosions, is common in OA. Different types of glenoid morphology are associated with shoulder OA, depending on the amount and localization of the glenoid erosion as well as the amount and direction of HHM. On the basis of these factors glenoids are classified in A, B, C and D types 4. In this classification A glenoid is a centered or symmetric arthritis without posterior subluxation of the humeral head. The B glenoid is characterized by asymmetric bone erosion, leading to glenoid retroversion, combined with posterior HHM. The D glenoid is defined by glenoid anteversion or anterior humeral head subluxation, while C glenoid is a dysplastic glenoid with at least 25° of retroversion "not caused by erosion.

Total shoulder arthroplasty (TSA) has been shown to relieve the pain and improve joint function of patients with OA. However, several complications such as component loosening and polyethylene damage has been reported and it has been revealed that 7.3% of glenoids may show signs of asymptomatic radiographic loosening annually after primary anatomic TSA. Although, aberrant glenohumeral contact mechanics has been suggested to be one of the primary potential causes, the mechanism of such fixation failure is still unclear. Glenohumeral conformity, eccentric loads associated with shoulder instability, bone quality, cementing techniques, implant orientation and design are all confounding factors that indeed affect the mechanical environment of the glenoid component, and, more specifically, also in terms of the contact mechanics.

Knowledge of in vivo glenohumeral joint contact mechanics before and after total shoulder arthroplasty and its interplay with patient- and surgery-related parameters may unravel the high rate of glenoid component loosening in patients with osteoarthritic glenoids and provide insight for the improvement of patient function, implant designs, implant longevity, and surgical technique. Previous ex-vivo and computational modelling studies that focused on the glenohumeral contact area after TSA, suggested that arm elevation in the scapular plane results in aberrant posterior translation of the humeral head in TSA patients. However, an in-vivo study based on dual-plane fluoroscopy, demonstrated that this only occurs in 50% of TSA patients. These discrepancies could arise from analyzing an assorted population of TSA patients without taking into account any specific information with regards to their preoperative osseous and soft-tissue status such as type of glenoid erosion, degree of glenoid retroversion, and amount of rotator cuff degeneration. Postoperative factors such as degree of retroversion correction, amount of joint-line medialization and glenohumeral components' radial mismatch were also not considered in these studies.

The main goal of this study is evaluating in-vivo glenohumeral contact patterns in patients with osteoarthritic glenoids before and after TSA, to unravel the high rate of glenoid component loosening. To that aim, the project is divided into four sub-objectives. The first objective is to compare glenohumeral contact areas before and after surgery in patients with osteoarthritic glenoids, using EOS (micro-dose x-ray) stereo radiographic imaging, to evaluate whether osseous correction during surgery is able to correct glenohumeral joint kinematics. The second objective is to compare OA patient's glenohumeral contact areas before and after surgery with healthy subjects. The third objective is to identifying variations in glenohumeral contact patterns after surgery with respect to the pre-and postoperative state of the patients. The last objective is to evaluate the influence of the location of the glenohumeral contact area after surgery on the long-term outcome and survival of the glenoid component.

ELIGIBILITY:
Inclusion Criteria:

OA patients group

* Patients with glenohumeral osteoarthritis planned for anatomic shoulder arthroplasty in the University Hospitals Leuven, Belgium
* Complete patient informed consent
* Pain free at the time of EOS imaging

Healthy control group

* Healthy adult volunteers with no history of shoulder pain or trauma
* Confirmation of the physician, that subject's clinical evaluation and CT scan did not show any abnormalities
* Complete informed consent

Exclusion Criteria:

Only patients with a functional TSA will be included, so patients with postoperative stiffness, pain, instability or pseudoparalysis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both OA patients and Healthy control group are screened in UZ Leuven
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Compere In-vivo glenohumeral joint contact patterns in patients using EOS stereo radiographic imaging | 2 years
  Evaluating in-vivo glenohumeral joint contact patterns in patients with different type of osteoarthritic glenoids pre- and post-TSA. Glenohumeral contact areas are compared before and after surgery in patients with osteoarthritic glenoids, using EOS stereo radiographic imaging
Compere in-vivo glenohumeral joint contact patterns in healthy subjects using EOS stereo radiographic imaging | 2 years
  Evaluating glenohumeral joint contact patterns in healthy subjects and comparing them with patients with osteoarthritic glenoids before patients receive surgery and after patients receive surgery. Glenohumeral contact areas are compared using EOS stereo radiographic imaging
Pre-operative factor: Humeral Head Migration | 2 years
  Identifying probable pre-operative factors; for example the amount of HHM; on glenohumeral contact area after surgery using pre- and postoperative CT scans.
Pre-operative factor: Inclination and rotator cuff muscle's quality | 2 years
  Identifying probable pre-operative factors; for example the inclination and rotator cuff muscle's quality; on glenohumeral contact area after surgery using pre- and postoperative CT scans.
Pre-operative factor: Degree of glenoid version | 2 years
  Identifying probable pre-operative factors; for example the degree of glenoid version; on glenohumeral contact area after surgery using pre- and postoperative CT scans.
Intra-operative factors: Degree of glenoid orientation correction | 2 years
  Identifying probable intra-operative factors; for example the degree of glenoid orientation correction; on glenohumeral contact area after surgery.
Intra-operative factors: Joint-line medialization | 2 years
  Identifying probable intra-operative factors; for example the joint-line medialization; on glenohumeral contact area after surgery.
Amount of osteolysis inside the glenoid vault and around glenoid component | 2 years
  Evaluating the amount of osteolysis inside the glenoid vault and around glenoid component of the patients at least 2 years after surgery

SECONDARY OUTCOMES:
Variations in glenohumeral contact areas | 2 years
  Determining possible variations in glenohumeral contact areas among patients with different type of osteoarthritic glenoids (A, B, C and D glenoids).
Influence of the location of the glenohumeral contact pattern | 2 years
  Evaluate the influence of the location of the glenohumeral contact area and amount of their deviations from healthy subjects on the long-term outcome and survival of the glenoid component. Pre-operative and 2 years after surgery, a CT scan from OA group will be obtained , which will be used for evaluating long-term outcome and survival of the glenoid component .

CONTACTS AND LOCATIONS:
Overall Officials: Filip Verhaegen, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided